CLINICAL TRIAL: NCT02654223
Title: Double Blind, Placebo-controlled, Dose Finding, Prospective, Multicenter Clinical Trial for the Treatment of Rhinitis/Rhinoconjunctivitis Against Grass Pollen Allergy
Brief Title: Dose Finding for the Treatment of Rhinitis/Rhinoconjunctivitis Against Grass Pollen Allergy
Acronym: MG56
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: MG56-SIT-012; 2014-005471-88 (EudraCT Number)
Record Dates: First submitted 2015-12-22; First posted 2016-01-13 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Rhinitis; Rhinoconjunctivitis
Keywords: Rhinitis / Rhinoconjunctivitis; Vaccine; Immunotherapy; Grass pollen; Allergy
MeSH Terms: conditions — Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- MG56 Mannosylated 500 subcutaneous (Experimental): 500 mTU/mL of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MG56 Mannosylated 500 subcutaneous; Biological: Sublingual placebo
- MG56 Mannosylated 1000 subcutaneous (Experimental): 1000 mTU/mL of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MG56 Mannosylated 1000 subcutaneous; Biological: Sublingual placebo
- MG56 Mannosylated 3000 subcutaneous (Experimental): 3000 mTU/mL of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MG56 Mannosylated 3000 subcutaneous; Biological: Sublingual placebo
- MG56 Mannosylated 5000 subcutaneous (Experimental): 5000 mTU/mL of subcutaneous immunotherapy and sublingual placebo.
  Interventions: Biological: MG56 Mannosylated 5000 subcutaneous; Biological: Sublingual placebo
- MG56 Mannosylated 500 sublingual (Experimental): 500 mTU/mL of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MG56 Mannosylated 500 sublingual; Biological: Subcutaneous placebo
- MG56 Mannosylated 1000 sublingual (Experimental): 1000 mTU/mL of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MG56 Mannosylated 1000 sublingual; Biological: Subcutaneous placebo
- MG56 Mannosylated 3000 sublingual (Experimental): 3000 mTU/mL of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MG56 Mannosylated 3000 sublingual; Biological: Subcutaneous placebo
- MG56 Mannosylated 5000 sublingual (Experimental): 5000 mTU/mL of sublingual immunotherapy and subcutaneous placebo.
  Interventions: Biological: MG56 Mannosylated 5000 sublingual; Biological: Subcutaneous placebo
- Placebo Sublingual Placebo subcutaneous (Placebo Comparator): Sublingual and subcutaneous placebo.
  Interventions: Biological: Subcutaneous placebo; Biological: Sublingual placebo

INTERVENTIONS:
Biological: MG56 Mannosylated 500 subcutaneous — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 500 mTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MG56 Mannosylated 500 subcutaneous
Biological: MG56 Mannosylated 1000 subcutaneous — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 1000 mTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MG56 Mannosylated 1000 subcutaneous
Biological: MG56 Mannosylated 3000 subcutaneous — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 3000 mTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MG56 Mannosylated 3000 subcutaneous
Biological: MG56 Mannosylated 5000 subcutaneous — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 5000 mTU (Mannosylated Therapeutic Units)/ml subcutaneous
  Arms: MG56 Mannosylated 5000 subcutaneous
Biological: MG56 Mannosylated 500 sublingual — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 500 mTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MG56 Mannosylated 500 sublingual
Biological: MG56 Mannosylated 1000 sublingual — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 1000 mTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MG56 Mannosylated 1000 sublingual
Biological: MG56 Mannosylated 3000 sublingual — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 3000 mTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MG56 Mannosylated 3000 sublingual
Biological: MG56 Mannosylated 5000 sublingual — Mixture of the following pollens: Phleum pratense, Dactylis glomerata, allergen extract with a concentration of 5000 mTU (Mannosylated Therapeutic Units)/ml sublingual
  Arms: MG56 Mannosylated 5000 sublingual
Biological: Subcutaneous placebo — Comparison between placebo and active group
  Arms: MG56 Mannosylated 1000 sublingual; MG56 Mannosylated 3000 sublingual; MG56 Mannosylated 500 sublingual; MG56 Mannosylated 5000 sublingual; Placebo Sublingual Placebo subcutaneous
Biological: Sublingual placebo — Comparison between placebo and active group
  Arms: MG56 Mannosylated 1000 subcutaneous; MG56 Mannosylated 3000 subcutaneous; MG56 Mannosylated 500 subcutaneous; MG56 Mannosylated 5000 subcutaneous; Placebo Sublingual Placebo subcutaneous

SUMMARY:
The purpose of the study is to evaluate the more efficient dose for the treatment of rhinitis/rhinoconjunctivitis against grass pollen allergy

DETAILED DESCRIPTION:
Double blind placebo-controlled study. The subjects will receive medication during 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Positive suggestive clinical history of intermittent or persistent moderate to severe rhinitis /rhinoconjunctivitis, with or without moderate asthma, due to grass pollen allergy
* Subjects with a positive skin prick-test (wheal sixe >6 mm diameter) Specific immunoglobulin E (IgE, CAP >3) to grass pollen
* Age between 14 and 65 years
* Both genders
* Subjects capable of giving informed consent
* Subjects capable of complying with the dosing regimen
* Subjects that have not received immunotherapy in the last 5 years
* Subjects presenting sensitization to another aeroallergens and or mites, cats or dogs, but that is considered clinically not relevant or no clinical interference with the nasal provocation test.

Exclusion Criteria:

* Subjects outside of the age range.
* Subjects who have previously received immunotherapy for the treatment of the allergic rhinitis/rhinoconjunctivitis due to grass pollen and other allergens in the last 5 years.
* Subjects that immunotherapy may be an absolute contraindication according to the criteria of the immunotherapy Committee of the Spanish society of Allergy and Clinical Immunology, and of the European Allergy and Clinical Immunology Immunotherapy Subcommittee may also include.
* Subjects with important symptoms of rhinoconjunctivitis /bronchial asthma in which the suspension of the systemic antihistamine treatment is contraindicated.
* Subjects with persistent severe or not controlled asthma , with a forced expiratory volume (FEV) < 70 respect to the reference value in spite of the appropriate pharmacological treatment at the time of the inclusion in the trial.
* Subjects that have required oral corticosteroids in the 12 weeks previous to the inclusion in the trial.
* Subjects that have previously submitted a serious secondary reaction during the skin prick test
* Subjects in treatment with beta blockers.
* Unstable subjects from the clinical point of view (respiratory infection, febrile, acute urticaria, etc.) at the time of the inclusion in the clinical trial
* Subject with chronic urticaria in the last 2 years or hereditary angioedema.
* Subjects that have some pathology (hyperthyroidism, hypertension, heart disease, etc.) is contraindicated.
* Subjects with any other disease not associated with the rhinitis/rhinoconjunctivitis, but of potential severity and that could interfere with treatment and follow-up (epilepsy, psychomotor deterioration, diabetes, malformations, multi-operated, kidney diseases,...).
* Subjects with autoimmune disease (lupus, thyroiditis, etc.), tumor or with diagnosis of immunodeficiency diseases.
* Subject whose status prevents him from providing cooperation and or which present severe psychiatric disorders.
* Subject with known allergy to other components of the vaccine different from pollen of grasses.
* Subjects with lower airway diseases other than asthma such as emphysema or bronchiectasis.
* Direct investigator's relatives.
* Pregnant or women at risk of pregnancy and breastfeeding women.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Concentration required to elicit a positive response after nasal provocation test (NPT) | 4 months
  Change in the threshold concentration of grass allergen extract, measured in Histamine Equivalent Prick per ml (HEP/ml), needed to trigger a positive response after nasal provocation test (NPT) assessed by acoustic rhinometry.
  This will be compared between the beginning and end of the trial and among active groups and placebo.

SECONDARY OUTCOMES:
Dose finding skin prick test | 4 months
  Comparison between the beginning and end of the trial and among active groups and placebo
Cytokine production by T cells specific allergen | 4 months
  Comparison between the beginning and end of the trial and among active groups and placebo
Immunoglobulin production by B cells specific allergen | 4 months
  Comparison between the beginning and end of the trial and among active groups and placebo
Phenotypic and functional analysis of dendritic cells | 4 months
  Will be analyzed changes in the frequency of plasmacytoid dendritic cells, myeloid dendritic cell and Treg cells in peripheral blood, between the beginning and end of the trial and among active groups and placebo
  The frequencies of peripheral blood mononuclear cells in each of the above populations is determined before and after treatment with mannosylated polymers by flow cytometry after staining with specific antibodies.
Number of participants with treatment-related adverse events as assessed by MG56-SIT-012 | 4 months
  Comparison between the beginning and end of the trial and among active groups and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Javier Subiza, PhD; MD, Principal Investigator — Clinica Subliza; Carmen Diéguez, PhD; MD, Principal Investigator — Hospital Universitario 12 de Octubre; Pedro Ojeda, PhD; MD, Study Director — Clínica Ojeda; Javier Ruiz Hornillos, PhD; MD, Principal Investigator — Hospital Universitario Infanta Elena; Matilde Domínguez, PhD; MD, Principal Investigator — Hospital Universitario Puerta de Hierro; Emilio Solano, MD, Principal Investigator — Hospital Universitario Ramón y Cajal; Antonio Moreno, Principal Investigator — Clínica Atlas; Pedro Guardia, Principal Investigator — Hospital Universitario Virgen Macarena; Agustín Orovigt, Principal Investigator — Hospital Viamed Santa Ángela de la Cruz; Alberto Caso, Principal Investigator — Hospital San Agustín; Alicia Alonso, Principal Investigator — Clínica Alianza Médica; Amparo Conde, Principal Investigator — Hospital Nisa Sevilla Aljarafe
Locations (12):
- Spain (12):
  - Clínica Atlas, Aranjuez, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - Hospital Nisa Aljarafe, Castilleja de la Cuesta, Sevilla
  - Hospital San Agustín, Dos Hermanas, Sevilla
  - CLÍNICA Dr. SUBIZA, Madrid
  - Clínica Ojeda, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - HOSPITAL UNIVERSITARIO 12 de OCTUBRE, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Viamed Santa Angola de la Cruz, Seville
  - Clínica Alianza Médica, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ojeda P, Barjau MC, Subiza J, Moreno A, Ojeda I, Solano E, Alonso A, Caballero R, Del Pozo S, Gomez-Perosanz M, Sanchez-Trincado JL, Benito-Villalvilla C, Angelina A, Soria I, Reche PA, Palomares O, Subiza JL, Casanovas M. Grass pollen allergoids conjugated with mannan for subcutaneous and sublingual immunotherapy: a dose-finding study. Front Immunol. 2024 Jun 26;15:1431351. doi: 10.3389/fimmu.2024.1431351. eCollection 2024. PMID 38989287